CLINICAL TRIAL: NCT03395834
Title: Comparison of Change of Tissue Oxygenation During a Vascular Occlusion Test Using Two Different Near-infrared Spectroscopy (O3TM vs. INVOS®)
Brief Title: Comparison of Change of Tissue Oxygenation During a Vascular Occlusion Test Using Two Different NIRS (O3TM vs. INVOS®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1712-054-905
Record Dates: First submitted 2017-12-24; First posted 2018-01-10 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Tissue Oxygen Saturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- O3 monitor (Experimental): tissue oxygenation comparison of O3 & INVOS
  Interventions: Device: O3

INTERVENTIONS:
Device: O3 — O3 TM and INVOS® monitoring simultaneously in single patient during 3 min of vascular occlusion test

SUMMARY:
This study evaluates the change of tissue oxygenation during a vascular occlusion test using two NIRS ( O3TM and INVOS®). NIRS probe will be attached on volunteer's forearm during vascular occlusion test and tissue oxygenation change will be recorded

DETAILED DESCRIPTION:
Near-infrared spectroscopy (NIRS) has been used to measure regional hemoglobin oxygen saturation of tissue. Recently, it also has been used to monitor peripheral tissue oxygen saturation, and micro-vascular reactivity using vascular occlusion test (VOT).

O3 TM is recently developed NIRS and there are only two clinical trials using this device, until now. In one study, this device could adequately predict cerebral regional oxygen saturation. And in the other study, peripheral tissue oxygenation was measured during ischemic pre-conditioning in heart surgery and it showed correlation between O3 TM and other NIRS ( EQUANOX) which has been used to monitor peripheral tissue oxygenation. But in this study, study group was patient with heart disease and the deoxygenation and reoxygenation rate during VOT was not not measured, which reflects tissue oxygen extraction and micro-vascular reactivity.

In NIRS devices, there are assumed cerebral arterial-venous ratio upon which oximetry values are calculated. In INVOS®, assumed arterial-venous ratio is 25/75. In other NIRS, assumed arterial-venous ratio is 30/70. But unlike other NIRS, O3 TM can change its preset arterial-venous ratio between 25/75 and 30/70, and there are no studies compare oximetry values between these two different settings.

In this study, the investigators try to compare INVOS®, which has been used widely for monitor tissue oxygenation, and two different settings of O3 TM ( arterial-venous ratio; 30/70 and 25/75). Three probes will be attached at same site simultaneously and the investigators will measure change of tissue oxygenation, deoxygenation rate and reoxygenation rate during vascular occlusion test

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult without known disease

Exclusion Criteria:

* Patients with previously known cardio-vascular disease
* Patients with body mass index >30kg/m2
* Patients on vasoactive drug
* Patients with skin pigmentation on probe attachment site
* Patients who is pregnant
* Patients with chronic anemia

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Change of tissue oxygenation during vascular occlusion test | stable baseline tissue oxygenation saturation ( less than 5 minutes) - 3 minute of vascular occlusion test - stable tissue oxygen saturation after reperfusion (less than 5 minutes)
  Change of tissue oxygenation measured by O3 (25/75), O3 (30/70) and INVOS® during vascular occlusion test

SECONDARY OUTCOMES:
deoxygenation rate (%/min) | stable baseline tissue oxygenation saturation ( less than 5 minutes) - 3 minute of vascular occlusion test - stable tissue oxygen saturation after reperfusion (less than 5 minutes)
  deoxygenation rate during vascular occlusion
reoxygenation rate (%/min) | stable baseline tissue oxygenation saturation ( less than 5 minutes) - 3 minute of vascular occlusion test - stable tissue oxygen saturation after reperfusion (less than 5 minutes)
  reoxygenation rate after reperfusion
Area under curve value of hyperemic area (% min) | stable baseline tissue oxygenation saturation ( less than 5 minutes) - 3 minute of vascular occlusion test - stable tissue oxygen saturation after reperfusion (less than 5 minutes)
  area under curve value of hyperemic area above baseline tissue oxygenation after reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University
Locations (3):
- South Korea (3):
  - SNUH, Seoul, Jongro Gu
  - Hee-Soo Kim, Seoul, Soul-t'ukpyolsi
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No